CLINICAL TRIAL: NCT03942835
Title: Psychometric Validation of the Competitive Attention Test (CAT) : Simultaneous and Separated Measures of Voluntary and Involuntary Attention
Brief Title: Psychometric Validation of the Competitive Attention Test
Acronym: CAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: abandonment
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0376; 2018-A02597-48 (Other: ID-RCB)
Record Dates: First submitted 2019-04-30; First posted 2019-05-08 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; attention; distraction; psychometric test; neuropsychological test validating procedure; psychostimulant
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy participants aged from 6 to 90 year-old (Experimental)
  Interventions: Other: experience 1 : Competitive attention test in healthy participants
- patients with ADHD with no treatment (Experimental): patients with ADHD aged from 6 to 90 year-old with no treatment
  Interventions: Other: experience 2 : Competitive attention test in patients with ADHD with no treatment
- patients with ADHD with treatment (Experimental): patients with ADHD aged from 6 to 90 year-old with psychostimulant treatment (Methylphenidate)
  Interventions: Other: experience 2 : Competitive attention test in patients with ADHD with no treatment; Other: experience 3 :Competitive attention test in patients with ADHD with psychostimulant treatment

INTERVENTIONS:
Other: experience 1 : Competitive attention test in healthy participants — Comparison of behavioral measures (reaction times and percentage of correct responses) obtained twice with the CAT test in healthy participants (2 to 6 weeks apart).
  Arms: Healthy participants aged from 6 to 90 year-old
Other: experience 2 : Competitive attention test in patients with ADHD with no treatment — Behavioral (reaction times and percentage of correct responses) and Electroencephalography (EEG) measures obtained with the CAT test in patients with ADHD with no treatment.
  Arms: patients with ADHD with no treatment; patients with ADHD with treatment
Other: experience 3 :Competitive attention test in patients with ADHD with psychostimulant treatment — Behavioral (reaction times and percentage of correct responses) and EEG measures obtained with the CAT test in patients with ADHD before and after psychostimulant treatment.
  Arms: patients with ADHD with treatment

SUMMARY:
This project aims at validating a new neuropsychological test to measure voluntary and involuntary attention for clinical use to diagnose attentional deficits.

This project proposes:

* a test-retest procedure in healthy subjects aged from 6 to 90 year-old;
* testing in attention deficit hyperactivity disorder (ADHD) patients before psychostimulant treatment;
* testing in attention deficit hyperactivity disorder (ADHD) patients before psychostimulant treatment.

ELIGIBILITY:
Inclusion Criteria:

healthy major participants:

* Age from 18 to 90 year-old
* Informed consent to participate in the study
* No neurological or psychiatric disorder
* No history of neuro-psychiatric disorder or neurodevelopmental type dysphasia, dyslexia, dyspraxia, attention deficit disorder

healthy minor participants:

* Age from 6 to 17 year-old
* Informed consent of parents or guardians for the child's participation in the study
* No neurological or psychiatric disorder
* No history of neuro-psychiatric disorder or neurodevelopmental type dysphasia, dyslexia, dyspraxia, Attention deficit disorder

ADHD minor patients:

* Age from 6 to 17 year-old
* Informed consent of parents or guardians for the child's participation in the study
* ADHD Diagnosis with or without hyperactivity
* No psychiatric history other than ADHD.
* For Experience 3: treatment in progress.

Exclusion Criteria:

healthy major participants

* Age below 18 or above 90 year-old
* unaffiliated or non-beneficiaries of the social security scheme

healthy minor participants:

* Age below 6 or above 18 year-old
* unaffiliated or non-beneficiaries of the social security scheme

ADHD minor patients:

* Age below 6 or above 18 year-old
* unaffiliated or non-beneficiaries of the social security scheme

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Reaction times in healthy subjects and patients with ADHD. | 6 weeks
  Reaction times in milliseconds obtained with the CAT test in healthy participants and in patients with ADHD.

SECONDARY OUTCOMES:
Percentage of correct responses in healthy subjects and patients with ADHD. | 6 weeks
  Percentage of correct responses obtained with the CAT test in healthy participants and in patients with ADHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Neurosciences de Lyon, INSERM U1028, Bron, France